CLINICAL TRIAL: NCT05079997
Title: Role of MAGNETIC RESONANCE IMAGING in Characterization of Superficial Soft Tissue Masses
Brief Title: MAGNETIC RESONANCE IMAGING in Superficial Soft Tissue Masses
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Alzahraa Mohamed Hassan Anwar, resident, Assiut University
Other Study IDs: mri in soft tissue
Record Dates: First submitted 2021-09-26; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Soft Tissue Masses
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MAGNETIC RESONANCE IMAGING — s a medical imaging technique used in radiology to form pictures of the anatomy and the physiological processes of the body. MRI scanners use strong magnetic fields, magnetic field gradients, and radio waves to generate images of the organs in the body. MRI does not involve X-rays or the use of ionizing radiation, which distinguishes it from CT and PET scans. MRI is a medical application of nuclear magnetic resonance (NMR) which can also be used for imaging in other NMR applications, such as NMR spectroscopy.

SUMMARY:
This study responds to these raise up questions: Can we use Diffusion Weighted MR complemented with numerical ADC values & in association with routine MRI in the discrimination between different malignant and benign superficial soft tissue masses.

DETAILED DESCRIPTION:
In the clinical practice, there is a large number & variety of superficial soft tissue masses. The differentiation of such masses represents a major obstacle for the surgeons. Benign &malignant neoplasms as well as non-neoplastic swellings may have similar clinical presentation. The differentiation between malignant & benign superficial soft tissue neoplasms is required for appropriate therapeutic planning and decisions. Masses can be characterized in terms of their size, number, component &vascularity using US and Doppler US. However, US is operator dependent & may display a number of artifacts that can result in misinterpretation. So MRI is superior in the assessment of such soft tissue masses due its brilliant soft tissue discrimination. Some features that will help distinguish malignant from benign lesions are evident on MRI examination such as signal characteristics,enhancement pattern,margin,lobulation,necrosis, haemorrhage,internal septation,peritumoral edema and extension through the deep fascia .However very forcful tumors may show benign behavior & appear similar to benign masses , Thus further histopathology is required for accurate diagnosis. Diffusion weighted MRI visualizes the random microscopic motion of molecules. Diffusion-weighted imaging (DWI) is the technique which allows measurement of the Brownian motion of water in the tissue microenvironment depending on the organization of the tissue, integrity of cell membranes, and tortuosity of extracellular space. Apparent Diffusion Coefficient (ADC) is a numerical parameter which is calculated from DWI. Previously, DWI technique was used with great success in the central nervous system (CNS), in the differentiation between benign and malignant tumors in addition to its great value in early diagnosis of recent strokes. Nowadays, DWI was used in the differentiation between malignant and benign soft tissue masses. Malignant tumors have abundant cellularity than benign tumors hence they have more restricted diffusion. The addition of quantitative ADC values plays a fundamental role in more accurate diagnosis of malignant superficial soft tissue neoplasms.

ELIGIBILITY:
Inclusion Criteria:

* patients with superficial soft tissue masses clinically
* patients underwent us detection of superficial soft tissue masses
* uncharactized superficial soft tissue mass by other modalities

Exclusion Criteria:

* MRI claustrophobia
* recurrent cases
* patients under treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with superficial soft tissue masses
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
benign and malignant masses | from october 2021 to october2022
  The discrimination between benign and malignant superficial soft tissue mass by Non invasive available technique

SECONDARY OUTCOMES:
Type of malignant superficial soft tissue masses | From October 2021 to October 2022
  Differentiation type of malignant superficial soft tissue masses

OTHER OUTCOMES:
Local invasion of malignant superficial soft tissue masses | From October 2021 to October 2022
  Detection local invasion of malignant superficial soft tissue masses

REFERENCES:
- [Background] Song Y, Yoon YC, Chong Y, Seo SW, Choi YL, Sohn I, Kim MJ. Diagnostic performance of conventional MRI parameters and apparent diffusion coefficient values in differentiating between benign and malignant soft-tissue tumours. Clin Radiol. 2017 Aug;72(8):691.e1-691.e10. doi: 10.1016/j.crad.2017.02.003. Epub 2017 Mar 6. PMID 28274509
- [Background] Thawait GK, Subhawong TK, Tatizawa Shiga NY, Fayad LM. "Cystic"-appearing soft tissue masses: what is the role of anatomic, functional, and metabolic MR imaging techniques in their characterization? J Magn Reson Imaging. 2014 Mar;39(3):504-11. doi: 10.1002/jmri.24314. Epub 2013 Oct 22. PMID 24532375
- [Background] Toprak H, Kilic E, Serter A, Kocakoc E, Ozgocmen S. Ultrasound and Doppler US in Evaluation of Superficial Soft-tissue Lesions. J Clin Imaging Sci. 2014 Feb 27;4:12. doi: 10.4103/2156-7514.127965. eCollection 2014. PMID 24744969
- [Background] Calleja M, Dimigen M, Saifuddin A. MRI of superficial soft tissue masses: analysis of features useful in distinguishing between benign and malignant lesions. Skeletal Radiol. 2012 Dec;41(12):1517-24. doi: 10.1007/s00256-012-1385-6. Epub 2012 Apr 12. PMID 22491777
- [Background] Herneth AM, Ringl H, Memarsadeghi M, Fueger B, Friedrich KM, Krestan C, Imhof H. Diffusion weighted imaging in osteoradiology. Top Magn Reson Imaging. 2007 Jun;18(3):203-12. doi: 10.1097/RMR.0b013e3180cac61d. PMID 17762384
- [Background] Panicek DM, Gatsonis C, Rosenthal DI, Seeger LL, Huvos AG, Moore SG, Caudry DJ, Palmer WE, McNeil BJ. CT and MR imaging in the local staging of primary malignant musculoskeletal neoplasms: Report of the Radiology Diagnostic Oncology Group. Radiology. 1997 Jan;202(1):237-46. doi: 10.1148/radiology.202.1.8988217.
- [Background] Fayad LM, Jacobs MA, Wang X, Carrino JA, Bluemke DA. Musculoskeletal tumors: how to use anatomic, functional, and metabolic MR techniques. Radiology. 2012 Nov;265(2):340-56. doi: 10.1148/radiol.12111740. PMID 23093707
- [Background] Kransdorf MJ, Murphey MD. Radiologic evaluation of soft-tissue masses: a current perspective. AJR Am J Roentgenol. 2000 Sep;175(3):575-87. doi: 10.2214/ajr.175.3.1750575. No abstract available. PMID 10954433
- [Background] Gielen JL, De Schepper AM, Vanhoenacker F, Parizel PM, Wang XL, Sciot R, Weyler J. Accuracy of MRI in characterization of soft tissue tumors and tumor-like lesions. A prospective study in 548 patients. Eur Radiol. 2004 Dec;14(12):2320-30. doi: 10.1007/s00330-004-2431-0. Epub 2004 Jul 29. PMID 15290067
- [Background] Kauppinen RA. Monitoring cytotoxic tumour treatment response by diffusion magnetic resonance imaging and proton spectroscopy. NMR Biomed. 2002 Feb;15(1):6-17. doi: 10.1002/nbm.742. PMID 11840548
- [Background] Baur A, Reiser MF. Diffusion-weighted imaging of the musculoskeletal system in humans. Skeletal Radiol. 2000 Oct;29(10):555-62. doi: 10.1007/s002560000243. PMID 11127677
- [Background] Szafer A, Zhong J, Gore JC. Theoretical model for water diffusion in tissues. Magn Reson Med. 1995 May;33(5):697-712. doi: 10.1002/mrm.1910330516. PMID 7596275
- [Background] Subhawong TK, Jacobs MA, Fayad LM. Insights into quantitative diffusion-weighted MRI for musculoskeletal tumor imaging. AJR Am J Roentgenol. 2014 Sep;203(3):560-72. doi: 10.2214/AJR.13.12165. PMID 25148158
- [Background] Padhani AR, Liu G, Koh DM, Chenevert TL, Thoeny HC, Takahara T, Dzik-Jurasz A, Ross BD, Van Cauteren M, Collins D, Hammoud DA, Rustin GJ, Taouli B, Choyke PL. Diffusion-weighted magnetic resonance imaging as a cancer biomarker: consensus and recommendations. Neoplasia. 2009 Feb;11(2):102-25. doi: 10.1593/neo.81328. PMID 19186405
- [Background] Ross BD, Moffat BA, Lawrence TS, Mukherji SK, Gebarski SS, Quint DJ, Johnson TD, Junck L, Robertson PL, Muraszko KM, Dong Q, Meyer CR, Bland PH, McConville P, Geng H, Rehemtulla A, Chenevert TL. Evaluation of cancer therapy using diffusion magnetic resonance imaging. Mol Cancer Ther. 2003 Jun;2(6):581-7. PMID 12813138
- [Background] Costa FM, Ferreira EC, Vianna EM. Diffusion-weighted magnetic resonance imaging for the evaluation of musculoskeletal tumors. Magn Reson Imaging Clin N Am. 2011 Feb;19(1):159-80. doi: 10.1016/j.mric.2010.10.007. PMID 21129640
- [Background] Gonzalez RG, Schaefer PW, Buonanno FS, Schwamm LH, Budzik RF, Rordorf G, Wang B, Sorensen AG, Koroshetz WJ. Diffusion-weighted MR imaging: diagnostic accuracy in patients imaged within 6 hours of stroke symptom onset. Radiology. 1999 Jan;210(1):155-62. doi: 10.1148/radiology.210.1.r99ja02155. PMID 9885601
- [Background] Nagata S, Nishimura H, Uchida M, Sakoda J, Tonan T, Hiraoka K, Nagata K, Akiba J, Abe T, Hayabuchi N. Diffusion-weighted imaging of soft tissue tumors: usefulness of the apparent diffusion coefficient for differential diagnosis. Radiat Med. 2008 Jun;26(5):287-95. doi: 10.1007/s11604-008-0229-8. Epub 2008 Jul 27. PMID 18661213
- [Background] Maeda M, Matsumine A, Kato H, Kusuzaki K, Maier SE, Uchida A, Takeda K. Soft-tissue tumors evaluated by line-scan diffusion-weighted imaging: influence of myxoid matrix on the apparent diffusion coefficient. J Magn Reson Imaging. 2007 Jun;25(6):1199-204. doi: 10.1002/jmri.20931. PMID 17520732